CLINICAL TRIAL: NCT00897793
Title: A Pilot Study of TGF-beta as a Potential Target for Prevention of Radiation-Induced Injury
Brief Title: Growth Factor Levels in the Blood of Patients Undergoing Radiation Therapy for Epithelial Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC RAD 0576; P30CA068485 (NIH); VU-VICC-RAD-0576
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Lung Cancer; Prostate Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; limited stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; male breast cancer; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Breast Neoplasms, Male; Colonic Neoplasms; Rectal Neoplasms | interventions — Phlebotomy; Radiotherapy; X-Ray Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with epithelial cancers: Patients with head and neck cancer, and lung, breast, colorectal, and prostate cancers who are to undergo radiation therapy
  Interventions: Procedure: venipuncture; Radiation: radiation therapy

INTERVENTIONS:
Procedure: venipuncture — Venipuncture for blood samples. Samples will be tested for TGF-beta.
  Other Names: blood sample collection
Radiation: radiation therapy — Radiation treatments vary according to type of cancer and by patient per doctors' recommendation
  Other Names: x-ray treatment

SUMMARY:
RATIONALE: Measuring levels of transforming growth factor-beta (TGF-beta) in the blood of patients with epithelial cancers (head and neck, lung, breast, colorectal, and prostate) may help doctors predict how patients will respond to treatment with radiation therapy.

PURPOSE: This research study is measuring levels of TGF-beta in patients with epithelial cancers who are undergoing radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether there is a dose-dependent increase in TGF-beta following radiotherapy in patients with epithelial cancers.

OUTLINE: Patients undergo blood sample collection prior to treatment, 24-72 hours after the first fraction of radiotherapy, and at the end of radiotherapy. Patients will also be asked for a weekly blood sample, but this is optional. Samples are analyzed to compare pre- and post-treatment TGF-beta levels.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Known diagnosis of an epithelial cancer, including any of the following:

  * Head and neck
  * Lung
  * Breast
  * Colorectal
  * Prostate
* Radiotherapy must be a component of planned treatment therapy

PATIENT CHARACTERISTICS:

* No serious medical or psychiatric illnesses which would prevent informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have epithelial cancers and who will undergo radiation therapy
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
TGF-beta levels | day 1 prior to treatment, 24-72 hours after 1st treatment, weekly at treatment (optional) and at completion of treatment
  TGF-beta is a protein that can be detected in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee